CLINICAL TRIAL: NCT07090369
Title: Phase Ib Trial of 177Lu-PSMA-I&T Therapy in Combination With Olaparib and Pembrolizumab in Patients With Metastatic Castration Resistant Prostate Cancer
Acronym: LumOnate
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24/186
Record Dates: First submitted 2025-07-15; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Castrate Resistant Prostate Cancer (mCRPC)
Keywords: prostate cancer; olaparib; pembrolizumab; 177Lu-PSMA; metastatic castrate resistant prostate cancer; triplet therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — olaparib; BID protein, human; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 177Lu-PSMA + olaparib + pembrolizumab (Experimental): Patients will receive treatment in two parts. A cycle in both parts is 42 days.
  In part 1, patients will receive a combination of olaparib (oral; days 1-22), a fixed 7.4 GBq dose of 177Lu-PSMA (IV infusion; day 5) and pembrolizumab (IV infusion; days 1 and 22).
  In part 2, patients will be administered with single agent pembrolizumab (IV infusion; days 1 and 22) for an additional 12 cycles of treatment.
  Interventions: Drug: Olaparib (300 mg BID); Drug: Pembrolizumab; Radiation: 177Lu-PSMA-I&T

INTERVENTIONS:
Drug: Olaparib (300 mg BID) — oral tablet
Drug: Pembrolizumab — IV infusion
Radiation: 177Lu-PSMA-I&T — PSMA-I&T is a small molecule ligand that binds to the extra-cellular domain of the prostatespecific membrane antigen. PSMA-I&T is a small molecule ligand that binds to the extra-cellular domain of the prostatespecific membrane antigen

SUMMARY:
This phase 1b trial is designed to evaluate the safety and tolerability of olaparib in combination with 177Lutetium-Prostate Specific Membrane Antigen (177 Lu-PSMA) and pembrolizumab in patients with metastatic castration resistant prostate cancer (mCRPC).

DETAILED DESCRIPTION:
This phase 1b, multi-centre, single arm, open label study is designed to evaluate the safety and tolerability of olaparib in combination with 177Lu-PSMA with concurrent treatment with pembrolizumab in patients with mCRPC. Patients with mCRPC who have previously progressed an Androgen Receptor Pathway Inhibitor (e.g. enzalutamide, abiraterone, darolutamide/or apalutamide) and have not had prior exposure to anti-PD-1, anti-PD-L1/L2, anti-CD137, or anti-CTLA-4 antibody or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathway, platinums, PARP inhibitors or radionuclide therapy will be eligible for the study. Patients can have had prior exposure to docetaxel in the chemotherapy naïve setting or castrate setting.

This is a single arm study divided into two treatment parts. In Part 1, patients will receive olaparib (oral; day 1-22),177Lu-PSMA (IV infusion; day 5), and pembrolizumab (IV infusion; day 1 and 22) for a maximum of six cycles (cycle = 42 days) of treatment. In Part 2, patients will continue to be treated with single agent pembrolizumab (IV infusion; day 1 and 22) for a subsequent 12 cycles (cycle = 42 days) of treatment.

Patients will be followed up every six weeks after the last dose of treatment until disease progression by modified RECIST 1.1 and/or PCWG3, start of new anti-prostate cancer therapy, withdrawal of consent, death, or 2 years a er the last patient has commenced treatment, whichever is earlier.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have provided written informed consent using the LumOnate Patient Information and Consent Form (PICF)
2. Patient must be ≥ 18 years of age at Screening
3. Willing and able to comply with treatment schedule, laboratory testing, and other requirements of the study
4. Histologically confirmed adenocarcinoma of the prostate without neuroendocrine or small cell differentiation
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
6. At least 2 weeks since the completion of prior therapy, including surgery or radiotherapy
7. PSA > 5 ng/mL
8. Significant PSMA avidity on PSMA PET/CT, defined as a minimum uptake of SUVmax 15 at a site of disease, and SUVmax > 10 at other sites of disease ≥ 10mm (unless subject to factors explaining a lower uptake, e.g. respiratory motion, reconstruction artefact)
9. Radiographic evidence of metastatic disease documented with either bone scan or CT scan (Appendix 2)
10. Patients must have adequate bone marrow, hepatic and renal function documented within 28 days prior to registration, defined as:

    * Haemoglobin ≥ 100 g/L independent of transfusions (no red blood cell transfusion in last 8 weeks)
    * Absolute neutrophil count ≥ 1.5 x 109/L
    * Platelets ≥ 150 x 109/L
    * Total bilirubin ≤ 1.5 x upper limit of normal (ULN) except for patients with known Gilbert's syndrome
    * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x ULN if there is no evidence of liver metastasis or ≤ 5 x ULN in the presence of liver metastases
    * Albumin ≥ 30 g/L
    * Adequate renal function: Patients must have creatinine clearance (CrCl) estimated of ≥ 51 mL/min using the Cockcroft-Gault equation or based on a 24 hour urine test
11. Patients must have progressed on an ARPI (e.g. enzalutamide, abiraterone, darolutamide/or apalutamide). Determination of disease progression on an ARPI will be made by the local Investigator
12. Patients must have progressive disease defined as any one of the following:

    1. PSA progression: minimum of two rising PSA values from a baseline measurement with an interval of ≥ 1 week between each measurement. The PSA value at screening should be ≥ 5 ng/mL
    2. Soft tissue or visceral disease progression as per modified RECIST 1.1 criteria (Appendix 2)
    3. Bone progression: ≥ 2 new lesions on bone scan (Appendix 2)
13. Prior surgical orchiectomy or chemical castration maintained on ongoing luteinizing hormone-releasing hormone analogue (agonist or
14. Patients must have a life expectancy ≥ 24 weeks
15. Non-sterilised male patients who are sexually active with a female partner of childbearing potential must use a condom from screening to approximately 3 months after the last dose of treatment. Female partners of male patients should also use a highly effective form of contraception throughout this period
16. Patients who are deemed to have disease that is safe and amenable to biopsy based on screening PSMA PET scans will be mandated to consent to paired tumour biopsies at Screening and on treatment

Exclusion Criteria:

1. Prior chemotherapy for mCRPC. Prior docetaxel is permitted if given in the setting of hormone sensitive disease
2. Site(s) of disease that are FDG positive with low PSMA expression defined by PSMA SUVmax < 10
3. Extensive marrow disease defined by a "Super Scan" on bone scintigraphy or diffuse marrow infiltration on PSMA PET
4. Active brain metastases or leptomeningeal metastases
5. Any prior exposure to anti-PD-1, anti-PD-L1/L2, anti-CD137, or anti-CTLA-4 antibody or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathway
6. Any prior exposure to PARP inhibitors, platinum, or radionuclide therapy
7. Patients with a history or clinical features suggestive of myelodysplastic syndrome/acute myeloid leukaemia or previously known clonal haemopoiesis
8. Patients unable to swallow orally administered medications or with gastrointestinal disorders likely to interfere with the absorption of the study medication
9. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed Tomography scan or psychiatric illness/social situations that is likely to impede participation and /or compliance in the study
10. Patients with active, known, or suspected autoimmune disease Note: Patients with vitiligo, type 1 diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enrol
11. Patients with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 7 days of registration Note: Inhaled or topical steroids, and adrenal replacement doses > 10 mg daily prednisone are permitted in the absence of active autoimmune disease
12. Malignancy within the previous 2 years other than basal cell or squamous cell carcinomas, skin or melanoma in situ, or other cancers that are unlikely to recur within 24 months
13. Positive test for hepatitis B virus surface antigen (HBsAg) or hepatitis C ribonucleic acid (HCV PCR) indicating acute or chronic infection
14. Patients with symptomatic or impending cord compression unless appropriately treated beforehand and clinically stable
15. Persistent toxicities (CTCAE ≥ Grade 2) caused by previous cancer therapy, excluding alopecia
16. Previous history of interstitial lung disease or non-infectious pneumonitis
17. Resting ECG indicating uncontrolled, potentially reversible cardiac conditions, as judged by the Investigator (e.g., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, QTcF prolongation > 500 ms, electrolyte disturbances, etc.), or patients with congenital long QT syndrome
18. Known hypersensitivity to olaparib or pembrolizumab or any of the excipients of olaparib or pembrolizumab
19. Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV) 1/2. Only need to check this if there is a clinical history. HIV-infected (HIV1/2 antibody-positive) patients may participate if they meet all the following eligibility requirements:

    * They must be on an anti-retroviral regimen with evidence of at least two undetectable viral loads within the past 6 months on this same regimen; the most recent undetectable viral load must be within 12 weeks prior to registration
    * They must have a CD4 count ≥ 250 cells/µL over the past 6 months on this same anti-retroviral regimen and must not have had a CD4 count < 200 cells/µL over the past 2 years unless it was deemed related to the cancer and/or chemotherapyinduced bone marrow suppression
    * For patients who have received chemotherapy in the past 6 months, a CD4 count < 250 cells/µL during chemotherapy is permitted as long as viral loads were undetectable during this same chemotherapy
    * They must have an undetectable viral load and a CD4 count ≥ 250 cells/µL within 7 days prior to registration
    * They must not be currently receiving prophylactic therapy for an opportunistic infection and must not have had an opportunistic infection within 6 months prior to registration
20. Concomitant use of known strong cytochrome P450, family 3 (CYP3A) inhibitors (e.g., itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks
21. Concomitant use of known strong (e.g., phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (e.g. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for phenobarbital and enzalutamide, and 3 weeks for other agents
22. Previous allogenic bone marrow transplant or double umbilical cord blood transplantation
23. Participation in another clinical study with an investigational product or another systemic therapy administered within 3 weeks prior to registration

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 24 months from recruitment of last patient
  To describe the radiological progression free survival (modified RECIST 1.1 and/or PCWG3 criteria) of the combination of 177Lu-PSMA-I&T, olaparib and pembrolizumab
Safety of Combination Therapy | 24 months from recruitment of last patient
  To evaluate the safety of 177Lu-PSMA-I&T in combination with olaparib and pembrolizumab. All adverse events (AE's) will be reported using CTCAE 5.0, with the severity (grade) and causality (relationship to investigational products) recorded for each participant.

SECONDARY OUTCOMES:
PSA50 response rate | 24 months from recruitment of last patient
  To evaluate the PSA50 response rate
PSA90 response rate | 24 months from recruitment of last patient
  To evaluate the PSA90 response rate
PSA progression free survival | 24 months from recruitment of last patient
  To evaluate PSA progression free survival
Overall Survival | 24 months from recruitment of last patient
  To evaluate the overall survival
Objective Response Rates | 24 months from recruitment of last patient
  To evaluate objective response rates in patients with measurable disease by modified RECIST 1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No